CLINICAL TRIAL: NCT07255430
Title: Interaction Between Microbiome, Virome and Host Immunity Response in the Context of Protracted Bacterial Bronchitis
Brief Title: Airway Microbiome of Patients With Protracted Bacterial Bronchitis
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: BUN B3002025000069
Record Dates: First submitted 2025-10-01; First posted 2025-12-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Protracted Bacterial Bronchitis
Keywords: cough; Protracted Bacterial Bronchitis; microbiome
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Oropharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Protracted bacterial bronchitis diagnostic: Children under five years old who attend pediatric outpatient visits or well-child visits at University Hospital Antwerp (UZA) and are diagnosed with Protracted bacterial bronchitis.

SUMMARY:
This project aims to assess the relationship between the microbiome and virome composition, the immune responses, and the respiratory health of children with protracted bacterial bronchitis (PBB). In addition, we aim to evaluate how the standard treatment with azithromycin interacts with the components of the microbiome, virome and immune biomarkers.

DETAILED DESCRIPTION:
Protracted Bacterial Bronchitis (PBB) is an often underestimated disease, characterized by a persistent cough for more than four weeks, without other significant underlying symptoms. While generally treatable, it can lead to complications such as recurrent infections and airway damage (bronchiectasis). The reasons why some children develop PBB or subsequent complications while others do not remain unclear. Recent research suggests that an impaired immune response and microbiota dysbiosis may play a key role. This study aims to analyze the microbial and viral composition of the airways in children with PBB, its relationship with inflammation, and the effects of azithromycin. Oropharyngeal swabs will be collected from up to 160 children <5 years old diagnosed with PBB at UZA in a longitudinal setup during one year. At each routine consultation (five in total) and during an exacerbation episode, three oropharyngeal swabs will be collected from each child. The three swabs will be used to: (1) determine the microbiome composition using next-generation sequencing, (2) identify the virome composition using multiplex qPCR or similar approaches, and (3) quantify immune biomarkers (RNA and protein-level) and culture microbial isolates. These findings will help to better understand the role of the airway microbiome in young children with PBB and identify microorganisms that may have a pathogenic or protective role. Ultimately, this knowledge may contribute to the development of new and effective diagnostics and treatments for PBB from an early age.

ELIGIBILITY:
Inclusion Criteria:

* Children with PBB diagnosis according to case definition
* Consent form signed by parents or legal guardians

Exclusion Criteria:

* Comorbidities (HIV, asthma, chronic obstructive pulmonary disease, diabetes)
* Have had serious illnesses (meningitis, pneumonia, bacteremia, empyema, etc) in the previous three months, identified only at the time of enrollment.
* Have chronic respiratory conditions at the time of enrollment (non-PBB bronchiectasis not caused by PBB, CF, allergy, etc.).
* Having received mechanical ventilation.
* Having been hospitalized or used antibiotics in the previous three months at the time of enrollment.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under five years old diagnosed with PBB.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of respiratory microbiome composition | Baseline, 3 months, 6 months, 9 months, 12 months and during exacerbations
  Description: Analysis of microbiome communities in airway samples will be performed using amplicon or shotgun sequencing to determine relative microbial abundances (in percentages) as the unit of measure, coupled with the use of bioinformatic tools for community structure analysis.
Prevalence of respiratory viruses | Baseline, 3 months, 6 months, 9 months, 12 months and during exacerbations
  Description: Detection of respiratory viruses from airway samples using RT-qPCR. Unit of Measure: percentage of positive samples (in percentages).

SECONDARY OUTCOMES:
Immune biomarkers profiling in airway samples | Baseline, 3 months, 6 months, 9 months, 12 months and during exacerbations
  Immunological profiling will be performed in airway samples by determining (1) cytokine concentrations based on protein-level analysis such as ELISA (pg/mL) and/or (2) differential gene expression based on RNA analysis (log fold-change or similar metric).
Correlates of respiratory microbiome | Baseline, 3 months, 6 months, 9 months, 12 months and during exacerbations
  Description: Microbial profiles will be associated with demographic, epidemiological and clinical data collected through standardized questionnaires and clinical assessments to determine relevant correlates. Unit of Measure: Statistical association measure (e.g., correlation coefficients or similar).
Correlates of Protracted Bacterial Bronchitis | Baseline, 3 months, 6 months, 9 months, 12 months and during exacerbations
  PBB events will be associated with demographic, epidemiological and clinical data collected through standardized questionnaires and clinical assessments to determine relevant correlates. Unit of Measure: Effect estimates (odds/prevalence/hazard ratios or similar).

CONTACTS AND LOCATIONS:
Overall Officials: Kim Van Hoorenbeeck, Prof. dr., Principal Investigator — University Hospital, Antwerp; Irina Spacova, Prof. dr. ir., Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The metadata of participants in the study will be made available in a restricted access repository. For samples and data sharing, the researchers will work with the legal department to establish Material/Data Transfer Agreements. Sequencing data are available at the European Nucleotide Archive. Physical samples are their origin will be stored at the decentral hub of the Antwerp biobank.
Time Frame: After the completion of the study (intended in 2029) and before publication, sequences and related metadata will be deposited into the ENA database and made available indefinitely.
Access Criteria: After data deposition in ENA, the data will be publicly accessible to anyone using the ENA instructions https://www.ebi.ac.uk/ena/browser/downloading-data